CLINICAL TRIAL: NCT05136248
Title: Comparison of Ultrasound Guided Intra-articular Steroid Injection and Pericapsular Nerve Group Block (PENG) in Patients With Chronic Hip Pain
Brief Title: Comparison of the Effect of Intra Articular Steroid Injection and Pericapsular Nerve Group Block for Hip Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Selin Guven Kose, principal Investigator, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 84/18
Record Dates: First submitted 2021-09-30; First posted 2021-11-29 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Injections, Intra-Articular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intraarticular injection (Experimental): intra-articular steroid injection with the ultrasound guidance technique,
  Interventions: Procedure: intraarticular injection
- peng block (Active Comparator): Ultrasound guided drug injection between to iliopubic eminentia and psoas tendon
  Interventions: Procedure: peng block

INTERVENTIONS:
Procedure: intraarticular injection — Ultrasound-guided intraarticular injection
  Arms: intraarticular injection
Procedure: peng block — Ultrasound-guided PENG block
  Arms: peng block

SUMMARY:
The most common cause of hip joint dysfunction in the elderly is degenerative osteoarthritis of the hip. Innervation of the hip joint capsule is provided by the obturator nerve, the accessory obturator nerve, and the femoral nerve. With pericapsular nerve group block (PENG), by blocking the femoral nerve and the accessory obturator nerve, analgesia is successfully provided for the hip joint. Intra-articular injection of corticosteroids; It is used as an alternative to surgical interventions because it reduces inflammation and short-term pain and is a minimally invasive method. The investigators aim to compare and report patients who underwent ultrasound-guided intra-articular steroid injection and PENG block in terms of post-procedural pain scores and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Hip pain NRS > 4
* No pathologies in the laboratory and coagulation parameters

Exclusion Criteria:

* Rheumatological disease with hip involvement
* Systemic active infection
* Malignancy
* History of hip joint surgery
* History of traumatic hip injury
* Platelets values < 150.000 / µl
* History of bleeding disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-04-25 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
numerical rating scale (NRS) pain score | change from baseline to day 1, week 2, 4, 8 after the block
  The 11-point NRS consists of numbers between 0 and 10 where 0 indicates "no pain" and 10 indicates "maximum pain." The patient is instructed to identify one number between 0 and 10, which is best representative of their pain intensity.

SECONDARY OUTCOMES:
Quality of Life (WOMAC) | baseline to 8 weeks
  The Western Ontario and McMaster Universities (WOMAC) is a self-administered health status measure and consists of 24 items divided into three domains, which are pain, stiffness, and physical function, validated to patients with hip or knee osteoarthritis

OTHER OUTCOMES:
Change in Harris Hip Score (HHS) | baseline to 8 weeks
  The Harris Hip Score (HHS) is a joint-specific measure, and it consists of two sections: questions and a physical examination, including a range of motion and deformity items. The score has a maximum of 100 points with a maximum of 44 points for pain, 47 for function, 4 points for absence of deformity, and 5 points for a range of motion. The highest score of 100 points indicates the best function and no pain.

CONTACTS AND LOCATIONS:
Overall Officials: selin guven kose, Principal Investigator — Diskapi Teaching and Research Hospital
Locations (1):
- Diskapi Yildirim Beyazit Training and Research Hospital, Ankara, Turkey (Türkiye)